CLINICAL TRIAL: NCT05759104
Title: Treatment and Fate in Fistulizing Crohn's Disease in a Pediatric Population
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, CHABOT Caroline, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2022PI067
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Crohn Disease
Keywords: fistula; abscess; pediatrics; medical treatment; surgery; drug
MeSH Terms: conditions — Crohn Disease; Fistula; Abscess | interventions — Infliximab; Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Infliximab — Drug
  Other Names: Adalimumab; Ustékinumab
Procedure: Stomy — Surgery
  Other Names: Resection

SUMMARY:
Crohn's disease is a inflammatory bowel disease evolving towards the destruction of the intestinal wall resulting in stenosing or perforating complications (fistulas, abscesses).

The treatment of perforating Crohn's disease is not codified.

DETAILED DESCRIPTION:
The old dogmas leading to surgery after failure of medical treatment have recently been overturned, particularly since the advent of anti-TNFs.

Biotherapies now have a central place, including for complicated forms. Previous studies have already looked at the usefulness of anti-TNFs in stenosing forms, or concerning ano-perineal lesions, but what about digestive fistulas.

Indeed, data are scarce, especially in paediatrics.

ELIGIBILITY:
Inclusion Criteria:

* Minor patients (aged 3 to 18).
* Diagnosed with Crohn's disease.
* fistulizing crohn's disease

Exclusion Criteria:

- perianal crohn disease

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * In consultations or hospitalized.
  * CHRU and CHR of Lille, Strasbourg, Colmar, Besançon, Dijon, Reims and Nancy.
  * Over the period from January 2012 to January 2022.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
No fistula | 12 month
  Complete remission = clinical remission and biological remission and iconographic remission:
  * clinical remission (asymptomatic at 12 months from inclusion).
  * biological remission (normalization of biological parameters 12 months after inclusion).
  * iconographic remission (no active lesion, and in particular no visualized fistula)

IPD SHARING:
Plan to Share IPD: No